CLINICAL TRIAL: NCT03719690
Title: A 2 Cohort, Non-comparative, Pivotal Study Evaluating the Efficacy of Tipifarnib in Patients With Head and Neck Squamous Cell Carcinoma (HNSCC) With HRAS Mutations (AIM-HN) and the Impact of HRAS Mutations on Response to First Line Systemic Therapies for HNSCC (SEQ-HN)
Brief Title: Safety and Efficacy of Tipifarnib in Head and Neck Cancer With HRAS Mutations and Impact of HRAS on Response to Therapy
Acronym: AIM-HN/SEQ-HN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-007
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: HRAS Gene Mutation; HNSCC
Keywords: TIPIFARNIB; HEAD AND NECK CANCER
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AIM-HN (Experimental): Tipifarnib, Oral Tablet. Dose Level 1 orally, bid on days 1-7 and 15-21 of 28-day treatment cycles
  Interventions: Drug: Tipifarnib; Device: HRAS Detection Assay
- SEQ-HN (No Intervention): HNSCC patients in whom HRAS mutations were not identified (wild type HRAS HNSCC) and who consent to provide first line outcome data and additional follow up.

INTERVENTIONS:
Drug: Tipifarnib — Tablet for oral administration
  Arms: AIM-HN
Device: HRAS Detection Assay — In Vitro Assay to detect HRAS mutations
  Arms: AIM-HN

SUMMARY:
An international, multicenter, open-label, 2 cohort, non-comparative, pivotal study evaluating the efficacy of tipifarnib in HRAS mutant HNSCC (AIM-HN). The first cohort will assess the objective response rate (ORR) of tipifarnib in subjects with HNSCC with HRAS mutations. The second study cohort, SEQ-HN, is an observational sub-study including HNSCC patients in whom HRAS mutations were not identified (wild type HRAS HNSCC) and who consent to provide first line outcome data and additional follow up.

DETAILED DESCRIPTION:
KO-TIP-007 is an international, multicenter, open-label, 2 cohort, non-comparative, pivotal study evaluating the efficacy of tipifarnib in HRAS mutant HNSCC (AIM-HN) and the impact of HRAS mutations on response to first line systemic therapies for HNSCC (SEQ-HN). KO-TIP-007 has 2 study cohorts. The first study cohort, named AIM-HN, includes HNSCC subjects with HRAS mutations. AIM-HN subjects will receive treatment with tipifarnib and the outcome of this cohort will be evaluated for ORR by an independent review facility.

The second study cohort, SEQ-HN, is an observational sub-study including HNSCC patients in whom HRAS mutations were not identified (wild type HRAS HNSCC) and who consent to provide first line outcome data and additional follow up.

HNSCC patients in whom HRAS mutations are identified and who meet eligibility criteria will be offered participation in AIM-HN. HNSCC patients in whom HRAS mutations are not identified may participate in SEQ-HN only. These patients will be followed and the comparison of outcomes of HRAS mutant and HRAS wild type HNSCC will address the exploratory objective to determine the effect of HRAS mutation on the ORR of first line systemic therapy in patients with recurrent/metastatic HNSCC. Outcome data from subsequent lines of therapy will be collected.

ELIGIBILITY:
Inclusion Criteria:

AIM-HN

1. At least 18 years of age.
2. Histologically confirmed head and neck cancer (oral cavity, pharynx, larynx, sinonasal, nasopharyngeal, or unknown primary) of squamous histology not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
3. Documented treatment failure from most recent prior therapy (e.g. tumor progression, clinical deterioration, or recurrence), and from at least one prior platinum-containing regimen, in any treatment setting.
4. Known tumor missense HRAS mutation.
5. Measurable disease by RECIST v1.1.
6. ECOG performance status of 0-1.
7. Acceptable liver, renal and hematological function
8. Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

1. Histologically confirmed salivary gland, thyroid, (primary) cutaneous squamous or nonsquamous histologies (e.g. mucosal melanoma).
2. Received treatment for unstable angina within prior year, myocardial infarction within the prior year, cerebro-vascular attack within the prior year, history of New York Heart Association grade III or greater congestive heart failure, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
3. Non-tolerable Grade 2 or ≥ Grade 3 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
4. Active, uncontrolled bacterial, viral or fungal infections requiring systemic therapy. Known history of infection with human immunodeficiency virus or an active infection with hepatitis B or hepatitis C.
5. Received treatment for non-cancer related liver disease within prior year.
6. Other protocol defined exclusion criteria may apply

Inclusion Criteria: SEQ-HN

1. At least 18 years of age.
2. Histologically confirmed head and neck cancer (oral cavity, pharynx, larynx, sinonasal, nasopharyngeal, or unknown primary) of squamous histology.
3. Will or has received at least one systemic anti-cancer therapy for recurrent or metastatic HNSCC.
4. HRAS wildtype (i.e., have no identified tumor missense HRAS mutation).
5. Other protocol defined inclusion criteria may apply

Exclusion Criteria: SEQ-HN

1. Histologically confirmed salivary gland, thyroid, (primary) cutaneous squamous or nonsquamous histologies (e.g. mucosal melanoma).

5. Other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (29):
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - The Oncology Institute of Hope and Innovation - Anaheim, Whittier, California
  - Miami Cancer Institute, Miami, Florida
  - University of South Florida H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University Of Kansas Medical Center, Westwood, Kansas
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center-Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health San Antonio - Mays Cancer Center, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne
  - Royal North Shore Hospital, Saint Leonards
- Austria (2):
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Hanusch Krankenhaus Wiener Gebietskrankenkasse, Vienna
- Belgium (5):
  - Centre Hospitalier Universitaire Universite Catholique de Louvain Site Godinne, Yvoir, Namur
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Leuven, Leuven
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
- Germany (4):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Würzburg, Würzburg
- Greece (3):
  - University General Hospital of Athens Attikon, Chaïdári
  - University General Hospital of Larissa, Larissa
  - Bioclinic - Thessaloniki, Thessaloniki
- Italy (7):
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera S. Croce e Carle Cuneo, Cuneo
  - Ospedale Mater Salutis di Legnago, Legnago
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS - Istituto Nazionale dei Tumori - Milano, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Azienda Ospedaliera Universitaria Senese-L'ospedale Santa Maria alle Scotte, Siena
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Institut Kanser Negara, Putrajaya
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University Medical Centre, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (2):
  - Haukeland Universitetssjukehus, Bergen
  - Radiumhospitalet, Oslo
- South Korea (8):
  - National Cancer Center, Goyang-si
  - Chonbuk National University Hospital, Jeonju
  - Korea University Anam Hospital, Seoul
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (15):
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - HM Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Costa Del Sol, Marbella
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Hat Yai
- United Kingdom (6):
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 296 participants were enrolled (59 participants in AIM-HN and 237 participants in SEQ-HN) in 14 countries between March 2019 and May 2023.
Pre-assignment Details: This study consisted of 2 non-comparative sub-studies: (1) an interventional open-label, single-arm, pivotal study evaluating the efficacy of tipifarnib in mHRAS HNSCC (AIM-HN) and (2) an observational study to evaluate the impact of HRAS mutations on response to first line systemic therapies for HNSCC (SEQ-HN).
Groups:
- Tipifarnib Treatment Cohort: AIM-HN: Participants enrolled as part of AIM-HN received tipifarnib administered with food at a starting dose of 600 mg, orally, twice a day (bid) on Days 1-7 and 15-21 of 28-day cycles.
- Observational Cohort: SEQ-HN: Participants with HNSCC in whom HRAS mutations were not identified (wild type HRAS HNSCC) and who consented to provide first line outcome data and additional follow-up.
Period: Overall Study
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN | Observational Cohort: SEQ-HN
Started | 59 | 237
Safety Analysis Set (SAS) | 59 | 0
Modified Intent-to-Treat Analysis Set (mITT) | 59 | 0
Completed | 0 | 0
Not Completed | 59 | 237
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Death | 40 | 149
Not completed — Miscellaneous | 12 | 56
Not completed — Lost to Follow-up | 2 | 18
Not completed — Unwilling or unable to comply with study requirements | 0 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Tipifarnib Treatment Cohort: AIM-HN: Participants enrolled as part of AIM-HN received tipifarnib administered with food at a starting dose of 600 mg, orally, bid on Days 1-7 and 15-21 of 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN | Observational Cohort: SEQ-HN | Total
Number analyzed (Participants) | 59 | 237 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 144 | 175
  >=65 years | 28 | 93 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 59 | 74
  Male | 44 | 178 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 180 | 213
  Black or African American | 1 | 10 | 11
  Asian | 23 | 37 | 60
  American Indian or Alaska Native | 0 | 2 | 2
  Other | 2 | 7 | 9
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 8
  Not Hispanic or Latino | 55 | 217 | 272
  Not Reported | 3 | 9 | 12
  Unknown | 1 | 3 | 4
Variant Allele Frequency (VAF) Status [Count of Participants; unit: Participants] — Genetic testing was done for tumor tissue to confirm mutant (variant) allele frequency at Baseline. Population: Data collection and analysis of VAF status for participants in the Observational SEQ-HN Cohort was not pre-specified.
  Participants
    number analyzed (Participants) | 59 | 0 | 59
    Participants with low VAF (< 20%) | 9 |  | 9
    Participants with high VAF (>=20%) | 50 |  | 50

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in High Variable Allele Frequency (VAF) Population, as Assessed by Independent Review Facility (IRF)
Description: ORR was defined as the percentage of participants who experienced a best overall response (BOR) of complete response (CR; disappearance of all target lesions) or partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by IRF. 95% confidence interval (CI) was calculated by the exact binomial (Clopper-Pearson) method.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants with high VAF only. Data collection and analysis of ORR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 50
percentage of participants | 20.0 [10.03 to 33.72]

2. Secondary Outcome: ORR in All VAF Population, as Assessed by IRF
Description: ORR was defined as the percentage of participants who experienced a BOR of CR or PR and was assessed using RECIST v1.1 by IRF. 95% CI was calculated by the exact binomial (Clopper-Pearson) method.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants. Data collection and analysis of ORR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
percentage of participants | 18.6 [9.69 to 30.91]

3. Secondary Outcome: Duration of Response (DoR) in High VAF Population, as Assessed by IRF
Description: DoR was defined as the time from the date of first response (CR or PR [whichever occurred first]) to the date of progression of disease or death of any cause, whichever occurred first, in participants with a confirmed CR or PR and was assessed using RECIST v1.1 by IRF. Median was calculated using the Kaplan-Meier method. 95% CI was based on Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants with high VAF and available data only. Data collection and analysis of DoR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 10
months | 6.51 [3.877 to NA] — Upper CI was not reached due to lack of events.

4. Secondary Outcome: DoR in All VAF Population, as Assessed by IRF
Description: as for outcome 3
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants with available data. Data collection and analysis of DoR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 11
months | 6.51 [3.877 to NA] — Upper CI was not reached due to lack of events.

5. Secondary Outcome: Progression Free Survival (PFS) in High VAF Population, as Assessed by IRF
Description: PFS was defined as months from the first dose of the study drug to the first documented progressive disease (PD, appearance of one or more new lesions or at least a 20% increase in the sum of the diameters of target lesions) or death, whichever came first and was assessed using RECIST v1.1 by IRF. Median was calculated using the Kaplan-Meier method. 95% CI was based on Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants with high VAF and available data only. Data collection and analysis of PFS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 50
months | 2.60 [1.873 to 4.402]

6. Secondary Outcome: PFS in All VAF Population, as Assessed by IRF
Description: PFS was defined as months from the first dose of the study drug to the first documented PD or death, whichever came first and was assessed using RECIST v1.1 by IRF. Median was calculated using the Kaplan-Meier method. 95% CI was based on Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to 28 approximately months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants with available data. Data collection and analysis of PFS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
months | 2.23 [1.873 to 3.548]

7. Secondary Outcome: PFS Rate in High VAF Population, as Assessed by IRF
Description: PFS rate was defined as the percentage of participants who had not experienced documented PD or death, whichever came first and was assessed using RECIST v1.1 by IRF at 6 and 9 month timepoints. Percentage of participants was calculated using the Kaplan-Meier method. 95% CI was calculated using normal approximation to the log transformed cumulative hazard rate
Time Frame: 6 months and 9 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 50
percentage of participants
  6 months | 29 [16.2 to 42.9]
  9 months | 20 [8.9 to 33.6]

8. Secondary Outcome: PFS Rate in All VAF Population, as Assessed by IRF
Description: as for outcome 7
Time Frame: 6 months and 9 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants and available data. Data collection and analysis of PFS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
percentage of participants
  6 months | 26 [14.9 to 38.4]
  9 months | 18 [8.9 to 30.8]

9. Secondary Outcome: Overall Survival (OS) in High VAF Population
Description: OS was defined as months from first dose date until death from any cause. Median was calculated using the Kaplan-Meier method. 95% CI was based on Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants with high VAF only. Data collection and analysis of OS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 50
months | 6.97 [4.895 to 11.466]

10. Secondary Outcome: OS in All VAF Population
Description: as for outcome 9
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants. Data collection and analysis of OS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
months | 6.21 [4.370 to 9.035]

11. Secondary Outcome: OS Rate at 12 Months in High VAF Population
Description: OS rate was defined as the percentage of participants who had not experienced or death and was assessed at 12 months. Percentage of participants was calculated using the Kaplan-Meier method. 95% CI was calculated using normal approximation to the log transformed cumulative hazard rate.
Time Frame: 12 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 50
percentage of participants | 31 [17.2 to 46.6]

12. Secondary Outcome: OS Rate at 12 Months in All VAF Population
Description: as for outcome 11
Time Frame: 12 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
percentage of participants | 30 [17.2 to 43.7]

13. Secondary Outcome: Time to Response (TTR) in High VAF Population, as Assessed by IRF
Description: TTR was defined as months from treatment start to first CR or PR (whichever was first recorded) in participants with confirmed CR or PR and was assessed using RECIST v1.1 by IRF. TTR was summarized descriptively by summary statistics.
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants with high VAF and available data only. Data collection and analysis of TTR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (Full Range); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 10
months | 1.9 [1.7 to 3.8]

14. Secondary Outcome: TTR in All VAF Population, as Assessed by IRF
Description: as for outcome 13
Time Frame: Up to approximately 28 months
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for all VAF participants with available data. Data collection and analysis of TTR for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (Full Range); unit: months
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 11
months | 1.9 [1.7 to 18.4]

15. Secondary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) that started on or after the first dose of the study drug and within 30 days of the last administration of the study drug. Common Terminology Criteria for Adverse Events (CTCAE) v5.0 was used for toxicity grading (Grade 3: severe or disabling; Grade 4: life-threatening; Grade 5: death related to AE). Clinically significant changes in laboratory tests, vital signs, and electrocardiogram results were reported as AEs.
Time Frame: Up to approximately 28 months
Population: SAS: consisted of all participants in the AIM-HN who received at least one dose of tipifarnib. Analysis was pre-specified for participants in the AIM-HN Cohort only. Data collection and analysis of safety for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 59
Participants
  Any TEAEs | 58
  Any Grade 3 or Higher TEAEs | 43

16. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module 35 (EORTC QLQ-H&N35) Subscales
Description: Change from Baseline score in pain, swallowing, speech problems, and senses problems subscales of EORTC QLQ-H&N35 are summarized individually. Raw scores for each subscale were linear transformations and standardized to range (0 - 100), with higher scores representing worse levels of symptoms. Change from Baseline was calculated as End of Treatment Observed - Baseline with a negative change representing a reduction in symptoms.
Time Frame: Baseline and End of Treatment Visit (up to approximately 28 months)
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants in the AIM-HN Cohort with available data. Data collection and analysis of EORTC QLQ-H&N35 for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 27
score on a scale
  Pain | 0.0 [-41.7 to 58.3]
  Swallowing: number analyzed (Participants) | 26
  Swallowing | 8.3 [-58.3 to 75.0]
  Senses problems | 0.0 [-50.0 to 66.7]
  Speech problems: number analyzed (Participants) | 26
  Speech problems | 0.0 [-44.4 to 66.7]

17. Secondary Outcome: Change From Baseline in the EuroQol-Visual Analog Scale (EQ-VAS) Score
Description: The EQ-VAS forms part of the EQ-5D-5L and collects the self-rating health status from 0 (the worst imaginable health) to 100 (the best imaginable health). Change from Baseline was calculated as End of Treatment Observed - Baseline with a negative change representing an increase in symptoms.
Time Frame: Baseline and End of Treatment Visit (up to approximately 28 months)
Population: mITT Analysis Set: consisted of all participants who received at least one dose of tipifarnib. Analysis was pre-specified for participants in the AIM-HN Cohort with available data. Data collection and analysis of EQ-VAS for participants in the Observational SEQ-HN Cohort was not pre-specified.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN
Number analyzed (Participants) | 26
score on a scale | 3.5 [-30.0 to 60.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 28 months
Description: All-cause mortality - all enrolled participants. Serious AEs and other AEs - SAS: consisted of all participants in the AIM-HN who received at least one dose of tipifarnib. Analysis was pre-specified for participants in the AIM-HN Cohort only. Data collection and analysis of AEs for participants in the Observational SEQ-HN Cohort was not pre-specified.
Arm/Group | Tipifarnib Treatment Cohort: AIM-HN | Observational Cohort: SEQ-HN
All-Cause Mortality (participants affected / at risk) | 41/59 | 149/237
Serious Adverse Events (participants affected / at risk) | 28/59 | 0/0
Other Adverse Events (participants affected / at risk) | 56/59 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipifarnib Treatment Cohort: AIM-HN (N=59) | Observational Cohort: SEQ-HN (N=0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | NA
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Fatigue (General disorders) | 1 | NA
Sudden death (General disorders) | 1 | NA
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Mental status changes (Psychiatric disorders) | 1 | NA
Blood creatinine increased (Investigations) | 1 | NA
Head injury (Injury, poisoning and procedural complications) | 1 | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | NA
Atrial fibrillation (Cardiac disorders) | 1 | NA
Cardiac arrest (Cardiac disorders) | 1 | NA
Syncope (Nervous system disorders) | 1 | NA
Anaemia (Blood and lymphatic system disorders) | 4 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | NA
Pancytopenia (Blood and lymphatic system disorders) | 1 | NA
Dysphagia (Gastrointestinal disorders) | 1 | NA
Ileus (Gastrointestinal disorders) | 1 | NA
Melaena (Gastrointestinal disorders) | 1 | NA
Oesophageal stenosis (Gastrointestinal disorders) | 1 | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | NA
Rectal prolapse (Gastrointestinal disorders) | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 2 | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Pneumonia (Infections and infestations) | 9 | NA
Sepsis (Infections and infestations) | 3 | NA
Septic shock (Infections and infestations) | 2 | NA
Bacteraemia (Infections and infestations) | 1 | NA
Corona virus infection (Infections and infestations) | 1 | NA
Diverticulitis (Infections and infestations) | 1 | NA
Lung infection (Infections and infestations) | 1 | NA
Pneumonia Escherichia (Infections and infestations) | 1 | NA
Soft tissue infection (Infections and infestations) | 1 | NA
Staphylococcal bacteraemia (Infections and infestations) | 1 | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipifarnib Treatment Cohort: AIM-HN (N=59) | Observational Cohort: SEQ-HN (N=0)
Hypertension (Vascular disorders) | 5 | NA
Fatigue (General disorders) | 19 | NA
Asthenia (General disorders) | 6 | NA
Mucosal inflammation (General disorders) | 5 | NA
Pyrexia (General disorders) | 4 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Insomnia (Psychiatric disorders) | 8 | NA
Anxiety (Psychiatric disorders) | 3 | NA
Confusional state (Psychiatric disorders) | 3 | NA
Blood creatinine increased (Investigations) | 10 | NA
Weight decreased (Investigations) | 7 | NA
Alanine aminotransferase increased (Investigations) | 5 | NA
Aspartate aminotransferase increased (Investigations) | 4 | NA
Blood alkaline phosphatase increased (Investigations) | 4 | NA
Tachycardia (Cardiac disorders) | 4 | NA
Headache (Nervous system disorders) | 4 | NA
Dizziness (Nervous system disorders) | 3 | NA
Anaemia (Blood and lymphatic system disorders) | 29 | NA
Neutropenia (Blood and lymphatic system disorders) | 20 | NA
Leukopenia (Blood and lymphatic system disorders) | 13 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | NA
Lymphopenia (Blood and lymphatic system disorders) | 6 | NA
Nausea (Gastrointestinal disorders) | 16 | NA
Vomiting (Gastrointestinal disorders) | 13 | NA
Constipation (Gastrointestinal disorders) | 11 | NA
Diarrhoea (Gastrointestinal disorders) | 10 | NA
Dysphagia (Gastrointestinal disorders) | 5 | NA
Abdominal pain (Gastrointestinal disorders) | 4 | NA
Abdominal distension (Gastrointestinal disorders) | 3 | NA
Abdominal pain upper (Gastrointestinal disorders) | 3 | NA
Dry mouth (Gastrointestinal disorders) | 3 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | NA
Rash (Skin and subcutaneous tissue disorders) | 3 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | NA
Corona virus infection (Infections and infestations) | 3 | NA
Decreased appetite (Metabolism and nutrition disorders) | 12 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 9 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 6 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements in place between clinical trial sites and the Sponsor (or its agents) that govern discussion or publication of trial results by the sites or their employees after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03719690/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03719690/SAP_001.pdf